CLINICAL TRIAL: NCT02386709
Title: Study Evaluating the Utility of 18F-FDG PET in Assessing Early Response to Neoadjuvant Treatment in Patients With Mammary Gland Cancer
Brief Title: Study Evaluating the Utility of 18F-FDG PET in Assessing Early Response to Neoadjuvant Chemotherapy in Patients With Mammary Gland Cancer
Acronym: TREN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A000357-40
Record Dates: First submitted 2015-02-13; First posted 2015-03-12 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: FDG PET

ARMS (1):
- Experimental Arm (Experimental): 1. Diagnostic
  2. PET1 : before the neoadjuvant treatment
  3. start neoadjuvant treatment
  4. PET2: two weeks after the start of the first course of chemotherapy
  5. surgery
  Interventions: Device: FDG PET

INTERVENTIONS:
Device: FDG PET — FDG PET1 before neoadjuvant chemotherapy FDG PET2 after one cycle of neoadjuvant chemotherapy

SUMMARY:
Neoadjuvant chemotherapy is frequently proposed to patients with mammary gland cancer. The aim is to reduce tumor volume before surgical therapy. Obtaining a pathologic Complete Response (pCR) is regarded as a good prognostic factor with less risk of recurrence. The rate of pCR is about 20%, although there are important variations according to tumor subtype and the type of treatment. The objective of the new therapeutic strategies is to increase this response rate.

The purpose of this study is to investigate the possibility of early evaluation of neoadjuvant chemotherapy response after one cycle of neoadjuvant chemotherapy by positron emission tomography (PET) with (18) F-fluorodeoxyglucose (FDG) in patients.

ELIGIBILITY:
Inclusion Criteria:

* patient having been informed of the study
* patient affiliated to a social health insurance
* ≥ 18 years
* patient presenting a breast cancer histologically confirmed
* indication of neoadjuvant chemotherapy treatment (classification UICC: II or III)
* patient agrees with exploitation of his clinical, biological and image data

Exclusion Criteria:

* distant metastasis
* contraindications to chemotherapy
* contraindications to surgery
* refusal
* serious illness not balanced, subjacent infection
* pregnancy or breast feeding
* diabetes not controlled (glycemia> 8 mmol/L)
* psychiatric disease
* patient under supervision, trusteeship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2015-03-25 (Actual); Primary Completion 2028-03-25 (Estimated); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
difference of Δ SUV (Standardised Uptak Value) between 18F-FDG PET 1 and 18F-FDG PET2 to predict pCR during neoadjuvant chemotherapy | early metabolic response mesure by 18F-FDG PET (difference of Δ SUV) at 3 weeks after neoadjuvant chemotherapy to predict pathologic Complete Response (pCR) by exploiting PET data realized before treatment (PET1) and after a cure of chemothrapy (PET2)

SECONDARY OUTCOMES:
Δ SUV (Standardised Uptak Value) threshold at 3 weeks | Δ SUV threshold at 3 weeks allowing to show the absence of response to treatment
Progression free survival | relation between early metabolic response (difference of Δ SUV ) assessed by 18F-FDG PET at 3 weeks and Progression-free survival
modification of tumor perfusion by 18F-FDG PET | modifications of tumor perfusion befoire and after one cycle(3 weeks) neoadjuvant chemotherapy by exploiting PET/PDG data (PET1 and PET2)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre COCHET, MD, Principal Investigator — Centre Feores François Lelcerc
Locations (1):
- Emilie REDERSTORFF, Dijon, France